CLINICAL TRIAL: NCT02748265
Title: A Pilot Study of the Effects of Nebulized Epoprostenol (Flolan) and Systemic Phenylephrine on Arterial Oxygenation During One Lung Ventilation
Brief Title: Nebulized Epoprostenol (FLOLAN) and Phenylephrine on One Lung Ventilation (OLV)
Acronym: FLOLAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-7520
Record Dates: First submitted 2016-03-23; First posted 2016-04-22 (Estimated); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Oxygenation During One Lung Ventilation
MeSH Terms: interventions — Phenylephrine; Epoprostenol; Sevoflurane; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inhaled Epoprostenol, phenylephrine, sevoflurane (Other): Inhaled Epoprostenol (Flolan), phenylephrine, volatile anesthesia maintenance (Sevoflurane)
  Interventions: Drug: Inhaled Epoprostenol and phenylephrine; Drug: Sevoflurane
- Inhaled Epoprostenol phenylephrine & Propofol (Other): Inhaled Epoprostenol (Flolan), phenylephrine and intravenous anesthesia maintenance (Propofol)
  Interventions: Drug: Inhaled Epoprostenol and phenylephrine; Drug: Propofol

INTERVENTIONS:
Drug: Inhaled Epoprostenol and phenylephrine — After 30 minutes of one-lung ventilation, Epoprostenol 50 ng/kg/min is administered via nebuliser in the anesthesia circuit with phenylephrine administered intravenously
  Other Names: Prostacyclin
Drug: Sevoflurane — Volatile maintenance anesthesia
  Arms: Inhaled Epoprostenol, phenylephrine, sevoflurane
Drug: Propofol — Intravenous maintenance anesthesia
  Arms: Inhaled Epoprostenol phenylephrine & Propofol

SUMMARY:
This is a pilot study of a new use of Epoprostenol via inhalation (Epoprostenol is approved for intravenous use). The purpose of this study is to administered inhaled Epoprostenol and intravenous Phenylephrine to improve arterial oxygen tension during one-lung anesthesia either with volatile anesthesia (Sevoflurane) or with intravenous anesthesia (Propofol).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing esophagectomy via video assisted thoracoscopy surgery or open thoracotomy.
* Patients greater than eighteen years old that have the capacity to provide consent.
* Patients who weigh 89kg or less.
* Patients with a preoperative platelet count > 100,000mm3

Exclusion Criteria:

* Contraindication or allergy to any of the study drugs e.g. epoprostenol, phenylephrine, sevoflurane or propofol.
* Spirometry: Force expiratory Volume (FEV1) less than 80% predicted for age. Patients with spirometry indicative of obstructive lung disease are less likely to develop hypoxemia during OLV compared to patients with normal spirometry . These patients are likely to have a smaller treatment effect if any.
* A history of a bleeding diathesis.
* Use of a platelet inhibitor within the last seven days e.g. Aspirin, clopidogrel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Increase of arterial oxygen tension in mmHg, during one-lung ventilation surgery, in response to combined nebulized epoprostenol/phenylephrine treatment | Changes measured during surgery, from start of treatment at 30 minutes after one-lung ventilation (T30) to end of the 30 minutes treatment (T60).

SECONDARY OUTCOMES:
Changes in base status in pH | Changes measured during surgery, from start of treatment at 30 minutes after one-lung ventilation (T30) to end of the 30 minutes treatment (T60).
Differences between anesthetic technique -volatile vs. intravenous- in increase of arterial oxygen tension in mmHg, during one-lung ventilation surgery, in response to combined nebulized epoprostenol/phenylephrine treatment | Changes measured during surgery, from start of treatment at 30 minutes after one-lung ventilation (T30) to end of the 30 minutes treatment (T60).
Changes in mean arterial blood pressure in mmHg | Changes measured during surgery, from start of treatment at 30 minutes after one-lung ventilation (T30) to end of the 30 minutes treatment (T60).
Changes in platelet function count | Changes measured during surgery, from start of treatment at 30 minutes after one-lung ventilation (T30) to end of the 30 minutes treatment (T60).
Changes in acid status in pH | Changes measured during surgery, from start of treatment at 30 minutes after one-lung ventilation (T30) to end of the 30 minutes treatment (T60).

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hospital, 200 Elizabeth St., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No